CLINICAL TRIAL: NCT03831113
Title: Pharmacologically-based Strategies for Opioid Substitution Therapy During Pregnancy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Steve N. Caritis, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Steve N. Caritis, MD, Professor, Department of OB/Gyn/RS, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100128; R01HD096796 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-02-05 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Opiate Addiction; Pregnancy
Keywords: Buprenorphine; medication-assisted treatment (MAT) programs
MeSH Terms: conditions — Opioid-Related Disorders; Short Stature, Auditory Canal Atresia, Mandibular Hypoplasia, Skeletal Abnormalities

STUDY DESIGN:
Intervention Model Description: dose reductions will alternate between 1 or 2 mg weekly (magnitude group) or 2 mg reductions every 1 or 2 weeks (frequency group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnitude Group (Active Comparator): Subjects will receive alternating reductions of 1 mg or 2 mg weekly.
  Interventions: Drug: Magnitude Group
- Frequency Group (Active Comparator): Subjects will receive dose reductions of 2 mg on alternating intervals of 1 and 2 weeks.
  Interventions: Drug: Frequency Group

INTERVENTIONS:
Drug: Magnitude Group — Dose reductions will alternate between 1mg or 2 mg weekly until the subject is no longer taking buprenorphine or is at the lowest tolerable dose.
  Other Names: magnitude
  Arms: Magnitude Group
Drug: Frequency Group — Dose reductions of 2 mg will occur alternate between once weekly to biweekly until the subject is no longer taking buprenorphine or is at the lowest tolerable dose.
  Other Names: frequency
  Arms: Frequency Group

SUMMARY:
This study is a pharmacodynamic study in pregnant women evaluating the relationship between buprenorphine concentration and outcome such as opioid withdrawal symptoms , NAS scores, neurodevelopmental and neuroanatomic outcomes. Strategies to reduce opioid exposure will be explored. There are 4 specific aims but only specific aim 4 is a clinical trial and reported here. In specific aim 4, eligible consenting women on buprenorphine in an MAT clinic will be assigned to 2 dose reduction regimens and their response to dose reduction will be measured using a visual analog scale.

DETAILED DESCRIPTION:
Opioid use has reached a staggering level and the associated deaths, neonatal consequences and economic impact are devastating. Buprenorphine and methadone are the two most commonly used medications for pregnant women in a Medication Assisted Treatment (MAT) program. Yet, the target concentration of these agents is not clearly identified. Furthermore, the relationship between drug exposure and adverse effects such as Neonatal Abstinence Syndrome and neurodevelopmental outcomes is unclear but contemporary thinking is that exposure (defined by maternal dose) is unrelated to adverse outcomes. The benefit of an MAT strategy is based on strong clinical data that demonstrates an improvement in perinatal outcomes in women participating in an MAT program. However, some women prefer to stop opioid medications entirely , but are not afforded this option in many MAT programs. The possibility that MAT is associated with some harms has received little attention but there are data that suggest that opioids adversely affect the fetal brain. If MAT is indeed associated with potential harms, then the option of Medically Supervised Withdrawal could be considered.

This study will assess two dose reduction strategies in a cohort of women who desire a reduction or elimination of their opioid exposure. The magnitude group will reduce the dose by either 1 or 2 mg weekly. The frequency group will reduce their dose by 2 mg alternately in one or 2 weeks

ELIGIBILITY:
Inclusion Criteria:

1. On a stable dosing regimen of BUP for at least 2 weeks as part of an established medication- assisted treatment (MAT) program.
2. Willingness to undergo supervised dose reduction
3. Subject willingness to be assigned to either the Magnitude, or Frequency group.
4. Single gestation between 14-30 weeks at the initiation of the dose reduction
5. On a BUP dose between 6- 24 mg daily (lower doses will not provide sufficient data points)
6. Willingness to have urine samples tested for drugs of abuse and blood samples tested for BUP+M concentrations during the Medical Supervised Withdrawal (MSW) clinic appointments
7. Willingness to attend weekly or biweekly MSW clinic appointments and to have daily contact via text messaging and to complete daily logs of sleep quality, withdrawal symptoms and symptoms of craving.
8. Willingness to attend psychosocial support meetings as needed.

Exclusion Criteria:

1. Current use of cocaine, heroin, benzodiazepines, barbiturates, phencyclidine (PCP), or opioids other than BUP.
2. Currently taking more than two mental health medications
3. Active moderately severe depression (PHQ-9 score ≥15 or suicidal ideation)
4. Current incarceration
5. Lack of a phone or transportation to and from clinic
6. Major fetal malformation
7. Mother with significant vaginal bleeding or serious medical or obstetrical complication that could adversely affect the study
8. Planned delivery at another institution
9. HIV or AIDS
10. Diagnosis of schizoaffective disorder or psychosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women who have been prescribed buprenorphine by a Medication Assisted Treatment (MAT) clinic.
Enrollment: 13 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Caritis, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Univerity of Pittsburgh Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - High Risk Obstetrical Consultants, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in two Medication Assisted Treatment clinics either in Pittsburgh or in Knoxville.Recruitment started on 4/13/2019 and ended on 12/22/2022. All participants at the Tennessee site were assigned to the frequency group
Groups:
- Magnitude Group: Subjects will alternately reduce dose by 1 mg/week then 2 mg/week. This will be repeated until the lowest tolerable dose is achieved. VAS scores during the 1 mg /week period will be recorded and compared to the VAS scores during the 2 mg/ week reduction.
- Frequency Group: Subjects will alternately reduce dose by 2 mg/week then 2 mg every 2 weeks. This will be repeated until the lowest tolerable dose is achieved. VAS scores during the 2 mg /week period will be recorded and compared to the VAS scores during the 2 mg every 2 week reduction.
Period: Overall Study
Arm/Group | Magnitude Group | Frequency Group
Started | 1 | 12
Completed | 1 | 1
Not Completed | 0 | 11
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Magnitude Group: Subjects will receive alternating reductions of 1 mg and then 2 mg weekly. Dose reductions will continue until the subject is no longer taking buprenorphine or is at the lowest tolerable dose.
- Frequency Group: Subjects will receive dose reductions of 2 mg on alternating intervals of 1 and 2 weeks. Dose reductions will continue until the subject is no longer taking buprenorphine or is at the lowest tolerable dose.
- Total: Total of all reporting groups
Arm/Group | Magnitude Group | Frequency Group | Total
Number analyzed (Participants) | 1 | 12 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (0) | 32.4 (6.1) | 31.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: protocol violations, drop outs and non-compliance led to non analysis of 11 subjects
  Participants
    number analyzed (Participants) | 1 | 1 | 2
    Female | 1 | 1 | 2
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: protocol violations, drop outs and non-compliance led to non analysis of 11 subjects
  Participants
    number analyzed (Participants) | 1 | 1 | 2
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 1 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: difference between analyzed vs recruited due to non- compliance , drop out or protocol violations
  Participants
    number analyzed (Participants) | 1 | 1 | 2
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 1 | 1 | 2
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Scores
Description: The VAS questionnaire consists of 4 questions related to cravings (0 = not at all to 10 = very much), withdrawal (0 = no symptoms to 10 = symptoms all day), sleep quality (0 = best to 10 = worst), and sleep duration (0 = longest ever to 10 = shortest ever). The 4 component questions are summed to provide a single VAS score for that day. The daily scores are averaged over the week or for two weeks depending on how often the dose was changed. The average VAS scores for each reduction regimen are averaged and compared to the alternative dosing group.
Time Frame: 36 weeks
Population: only those compliant with protocol were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Magnitude Group: Group had dose reduced alternately by 1 or 2 mg weekly
- Frequency Group: participants reduced their dose by 2 mg either weekly or biweekly
Arm/Group | Magnitude Group | Frequency Group
Number analyzed (Participants) | 1 | 1
score on a scale
  1 mg or 1 week cycle | 2.11 (.12) | .43 (.13)
  2 mg or 2 week cycle | 1.94 (.23) | .43 (.13)

ADVERSE EVENTS:
Time Frame: Participants were evaluated over the time from enrollment until delivery, generally 6 months
Description: There was an impossibly high rate of no compliance as 11 of the 13 recruited subjects were noncompliant and repeatedly violated the protocol
Groups:
- Magnitude Group: Subjects will receive alternating reductions of 1 mg and then 2 mg weekly. Reductions will repeat till dose=0 or at the lowest possible dose
- Frequency Group: Subjects will receive dose reductions of 2 mg on alternating intervals of 1 and 2 weeks. Reductions will repeat till dose=0 or at the lowest possible dose.
Arm/Group | Magnitude Group | Frequency Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/12
Other Adverse Events (participants affected / at risk) | 0/1 | 0/12

LIMITATIONS AND CAVEATS:
This portion of the study was terminated due to poor recruitment and poor compliance of recruited subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03831113/Prot_SAP_000.pdf